CLINICAL TRIAL: NCT03757598
Title: ePartogram Effectiveness Study: A Mixed Methods Quasi-experimental Study in Kisumu and Meru, Kenya.
Brief Title: ePartogram Effectiveness Study in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ePartogram Kenya
Record Dates: First submitted 2017-11-28; First posted 2018-11-29 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Obstetric Complication; Obstetric Labor Complications; Newborn Morbidity
Keywords: partograph, labor, birth, complications, newborn, Kenya
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Intervention Model Description: There are two study groups, each with 6 health facilities. All providers offering maternity care were trained in labor management practices and use of the partograph approved for national use in Kenya. In the intervention group only, providers were offered training and Android tablets to use the electronic partogram with clients. The 6-month intervention phase was simultaneous in both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paper Partograph (No Intervention): The comparison group used the standard WHO Standard Paper Partograph approved in Kenya to monitor labor. Copies of the partograph were made available to the facilities.
- ePartogram (Experimental): ePartogram use by skilled birth attendant providers in health facilities. The intervention arm used the novel ePartogram or electronic partogram. The interface was of the same WHO approved partograph on an Android tablet. There were reminders to spur provider actions and alerts that were programmed in an algorithm.
  Interventions: Other: ePartogram use

INTERVENTIONS:
Other: ePartogram use — Electronic partograph based on WHO standard paper partograph is given in Android tablet used by provider monitoring clients in labor. Providers had received training in using the ePartogram and ongoing trouble shooting.
  Arms: ePartogram

SUMMARY:
Quasi-experimental study to evaluate whether clinical care offered to clients was more appropriate and in line with WHO recommendations for care in normally progressing labor and in labor with complications, among providers using the novel intervention, ePartogram (an electronic version of the WHO paper partograph) vs. providers who offered care using the standard paper partograph, and whether fetal/newborn outcomes were improved among cases where partograph was used.

DETAILED DESCRIPTION:
The ePartogram is an electronic version of the WHO Partograph and is developed by Jhpiego. Seventy-eight clinical rules, programmed into the ePartogram, are based on global guidelines in the WHO manual "Managing complications in pregnancy and childbirth: a guide for midwives and doctors" and the expert opinion of Jhpiego physicians and nurse-midwives. The rules underwent a validation process by 65 expert skilled birth attendants (SBAs) (working in maternity wards of health facilities) from a variety of geographic and clinical settings affiliated with Jhpiego. In the ePartogram application ("app") that is put on an Android tablet computer, the clinical rules trigger "reminders" to SBAs to take a routine clinical measurement, such as fetal heart rate (every 30 minutes) or maternal temperature (every 2 hours). The rules also trigger "low-level" alarms indicating a measurement that falls in the abnormal range that could be cause for concern (i.e. meconium-stained liquor), and "high-level" alarms that could indicate need for immediate action (i.e. maternal systolic blood pressure ≥160 mm Hg).

Litwin et al. reported on the feasibility and acceptability of use of an electronic partogram in Zanzibar and concluded that health workers felt the ePartogram improved timeliness of care and supported decision making. Health workers quickly became competent and confident in using the tablet device and ePartogram application. This study in Kenya has an objective to evaluate whether providers' use of the ePartogram improves labor outcomes and labor management in health facilities. The study design is a quasi-experimental design evaluation comparing data collected at 6 intervention sites and 6 comparison sites with similar facility characteristics and in two regions of Kenya.

ELIGIBILITY:
Inclusion Criteria:

Facilities:

* In Kisumu or Meru
* BEmONC or CEmONC sites
* At least one SBA on duty in labor ward 24 hours per day
* Facility in-charge or in-charge of L&D ward available physically or remotely 24 hours per day
* Use WHO modified paper partograph
* Adequate supply of paper partographs and maternity registers
* Availability of reliable transportation for referrals (e.g. functional ambulance) 24 hours per day

Providers:

* Providers meeting the WHO definition of Skilled Birth Attendant (SBA) clinical provider working in care for laboring women who will be working at the facility during the study.
* Providers completing the three-day labor management training comprised of training on partograph use and management of normal labors and labor complications, according to WHO and Kenya MOH guidelines
* Intervention sites only: Providers passing the ePartogram post-training test will be asked to use the ePartogram during clinical care.

Exclusion Criteria:

Facilities:

* Facility not registered with MOH
* No SBA on duty in labor ward at any time during a 24 hour period
* No in-charge available at any time during a 24 hour period
* Dispensary health facilities that do not practice BEmONC

Providers:

* Providers not meeting the WHO definition of SBA
* Providers not completing the labor management training or (intervention sites only) not passing the ePartogram post-training test

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Percent of partographs showing fetal/newborn with a suboptimal fetal/newborn outcome | All partographs within the 6 month intervention period; the partograph is started in the active phase of labor - at 4 cm dilatation - and may last up to 12 hours
  Percent of partographs with a suboptimal fetal/newborn outcome (defined by presence of fresh stillbirth, newborn Apgar score of 5 or below at 1 minute, or Apgar score of 7 or below at 5 minutes or newborn resuscitation needed -- as recorded on the partograph by the health provider)

SECONDARY OUTCOMES:
Percent of partographs with a suboptimal maternal outcome | All partographs within the 6 month intervention period; the partograph is started in the active phase of labor - at 4 cm dilatation - and may last up to 12 hours
  Percent of partographs with a suboptimal maternal outcome (defined by presence of retained placenta, blood loss at greater to or equal to 500 ml, systolic blood pressure of less than 90 or greater than 140, diastolic blood pressure of less than 60 or more than 90, and pulse at less than 60 or greater than or equal to 100), as recorded by the provider on the partograph
Action recorded on partograph to maintain normal labor, among all partographs or partograms | Six-month intervention period
  To support the objective of supporting decision-making and actions to maintain normal labor, there were additional items added to both the paper partograph and the electronic partogram that providers answered by ticking off actions to maintain normal labor. These 5 actions were: encouraging ambulation, giving food, giving fluids, offering the position of choice, encouraging a companion to be present. This indicator refers to any of these actions, and among all partographs or partograms
Action recorded by the provider to address any sign of non-normalcy in labor, among all partographs or partograms | Six-month intervention period
  To support the objective of: Detection, decision-making and action to address deviations from normal labor and complications arising during labor. Seven actions included: providing oxygen, changing the position of the laboring woman in response to FHR abnormalities, checking for bleeding, consulting with a supervisor, and referring a client to another facility, inducing labor during the first stage, and conducting an episiotomy. The indicator is any action taken.
Fresh stillbirth and neonatal death <24 hours out of all births, according to aggregate monthly routine facility data | Six-month intervention period and six-month pre-intervention period
  Fresh stillbirth and neonatal death <24 hours out of all births, according to aggregate monthly routine facility data recorded on facility registers by providers and aggregated by facility records staff

CONTACTS AND LOCATIONS:
Overall Officials: Sanghvi Harshad, MD, Principal Investigator — Jhpiego
Locations (12):
- Kenya (12):
  - Ahero Hospital, Kisumu
  - Kisumu Hospital, Kisumu
  - Kombewa Health Center, Kisumu
  - Lumumba Health Center, Kisumu
  - Nyabondo Hospital, Kisumu
  - Nyakach Health Center, Kisumu
  - Maua Methodist Hospital, Meru
  - Meru Teaching and Referral Hospital, Meru
  - Mikinduri Health Center, Meru
  - Muthara Health Center, Meru
  - Mutuati Health Center, Meru
  - Nyambene Hospital, Meru

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan to share study data. An investigator can contact harshad.sanghvi@jhpiego.org with a request. Jhpiego is developing an open data sharing process.

REFERENCES:
- [Background] Managing complications in pregnancy and childbirth: a guide for midwives and doctors - 2nd ed. Editors: World Health Organization Publication date: 2017 Languages: English ISBN: 9789241565493
- [Background] Litwin LE, Maly C, Khamis AR, Hiner C, Zoungrana J, Mohamed K, Drake M, Machaku M, Njozi M, Muhsin SA, Kulindwa YK, Gomez PP. Use of an electronic Partograph: feasibility and acceptability study in Zanzibar, Tanzania. BMC Pregnancy Childbirth. 2018 May 9;18(1):147. doi: 10.1186/s12884-018-1760-y. PMID 29743032

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT03757598/Prot_SAP_000.pdf